CLINICAL TRIAL: NCT01789190
Title: Observational Study: Regular Physical Exercise Extends Honeymoon Phase in Type 1 Diabetes Subjects
Brief Title: Regular Physical Exercise Extends Honeymoon Phase in Type 1 Diabetes Subjects
Acronym: Honeymoon
Status: Terminated | Type: Observational
Why Stopped: The study has concluded normally
Sponsor: University Hospital A Coruña (Other)
Collaborators: Universidad Miguel Hernandez de Elche (Other); University of Alicante (Other)
Responsible Party: Principal Investigator, Enrique Roche, PhD, University Hospital A Coruña
Other Study IDs: PS09/01093
Record Dates: First submitted 2013-02-05; First posted 2013-02-11 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2013-02

CONDITIONS: Type 1 Diabetes; Physical Activity
Keywords: Honeymoon; Type 1 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Group S (sedentary): Group S included patients that did not perform any physical activity at the moment of onset, continuing with the same habits during the subsequent observational period.
- Group A (active): The inclusion criteria for group distribution took in account the principles of the American College of Sports Medicine, considering as active physical activity to practice a moderate-vigorous exercise during 1h, 5 days or more/week. In this context, a sedentary or less active person should be a person that practices any or less than 5h weekly

SUMMARY:
In diabetes, the honeymoon period is characterized by the presence of a functional reserve of β-cells that favours an adequate metabolic control and low insulin needs in order to control glycaemia. Therefore, the extension of this period could have evident benefits in diabetes management. The investigators aimed to study the influence of regular physical activity on the prolongation of the honeymoon period

DETAILED DESCRIPTION:
Observational study of two groups of type 1 diabetic patients from onset to a two-year period. One group exercised regularly (5 or more hours/week) before onset and continued doing so with the same regularity (group A). The second group either did not perform physical activity or did so sporadically (group S).

Consultations were initially performed on a weekly basis for the first month, then once a month for the remaining period. In each consultation, patients were asked about diet accomplishment, glycaemia monitoring, insulin injections and exercise performance. All individuals from group A declared to practice regularly intervallic routines, playing team sports (basketball for n=1 and soccer for n=6). Only one individual declared to perform aerobic exercise (long distance running and swimming). At the end of the first year a second blood sample was extracted in the same conditions from each individual to determine the same parameters. Exercise routine accomplishment and follow-up of diet and insulin injections was followed monthly during one more year. At the end of this period, the study was considered finished and the last blood extraction was performed in order to measure the same parameters. Other subjects were excluded because they were not capable to provide data required for study follow up.

ELIGIBILITY:
Inclusion Criteria:

* Undergo type 1 diabetes.
* To practice a moderate-vigorous exercise during 1h, 5 days or more/week before onset and continuing practicing for 2 more years for group A (active).
* To practice any or less than 5h weekly before and after onset for group S (sedentary).
* Capable to provide data and blood samples during follow up.

Exclusion Criteria:

- Not capable to provide data and blood samples required for study follow up.

Ages: 7 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 19 subjects from 26 with recent onset of type 1 diabetes completed the 2 years study in the Endocrinology Service of the University Hospital Complex of A Coruña (Spain).
  The mean age of group A was 21.9±4.2 years and included 8 individuals, 5 men and 3 women diagnosed at the moment of onset by hyperglycaemia + ketoacidosis (n=4), ketoacidosis (n=2) or hyperglycaemia (n=2). The mean age of group S was 23.3±2.2 years and included 11 individuals, 7 men and 4 women diagnosed at the moment of onset by hyperglycaemia + ketoacidosis (n=3), ketoacidosis (n=7) or hyperglycaemia (n=1).
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2011-01; Primary Completion 2013-01 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
We aimed to study the influence of regular physical activity on the prolongation of the honeymoon period in type 1 diabetic patients by determining circulating parameters. | 2 years
  Circulating parameters to assess diabetes management: HbA1c was determined by immunoanalysis. C-peptide was determined by radioimmunoassay using the Coat-a-Count kit (Diagnosis Products Corporation, LA). Protein carbonyl derivatives were calculated by adapting the method developed by Levine (1994) (12)

SECONDARY OUTCOMES:
To study the influence of regular physical activity on the control of the inflammation process associated to type 1 diabetes. | 2 years
  Inflammation was assessed by determining circulating cytokines were in plasma by Flow Cytometry (FACSCalibur, Benton & Dickinson Bioscience) through the FlowcytomixTM Multiplex Test (eBioscience) (n=3). The following cytokines were analysed for each patient: IL (interleukin)-1beta, IL-2, IL-4, IL-5, IL-6, IL-9, IL-10, IL-12p70, IL-13, IL-17a, IL-22, TNF (tumor necrosis factor)-alpha and INF (interpheron)-gamma.

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Martinez-Ramonde, MD, Principal Investigator — Endocrinology Departmente, Hospital A Coruna
Locations (1):
- Endocrinology Service of the University Hospital Complex of A Coruña (Spain), A Coruña, A Coruna, Spain

REFERENCES:
- See also: PDF of the study — https://sites.google.com/a/goumh.umh.es/clinicaltrials/anuncios